CLINICAL TRIAL: NCT00967551
Title: The Impact of the Use of Zinc Supplementation and Other Micronutrients on the Occurence of Diarrhea Diseases and Respiratory Infections in Children of Daycare Centers
Brief Title: Micronutrient Sprinkles in a Daycare Center
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Conrad R. Cole, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00007903
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Results first posted 2013-04-08 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Diarrhea; Respiratory Infection
Keywords: Diarrhea; Pneumonia; Upper respiratory infections; Acute gastroenteritis
MeSH Terms: conditions — Diarrhea; Respiratory Tract Infections; Pneumonia | interventions — Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Micronutrient Sprinkles without zinc (Active Comparator): Micronutrient sprinkles without zinc
  Interventions: Dietary Supplement: Micronutrient sprinkles without zinc
- Micronutrient sprinkles with zinc (Experimental): Micronutrient sprinkles with zinc gluconate
  Interventions: Dietary Supplement: Micronutrient Sprinkles with zinc

INTERVENTIONS:
Dietary Supplement: Micronutrient Sprinkles with zinc — Daily dose of 1 packet of sprinkles
  Other Names: Micronutrient sprinkles
  Arms: Micronutrient sprinkles with zinc
Dietary Supplement: Micronutrient sprinkles without zinc — I packet of micronutrient sprinkles without zinc
  Other Names: Micronutrient sprinkles
  Arms: Micronutrient Sprinkles without zinc

SUMMARY:
Diarrheal diseases are a major cause of morbidity and mortality globally in children less than 5 years of age. Prolonged diarrhea, recurrent infections and growth failure in developing countries are usually a consequence of micronutrient deficiencies including zinc. The primary aims of the proposed study are to evaluate the effect of the use of multiple micronutrient sprinkles including zinc on compliance of supplement use and the incidence of recurrent diarrheal and respiratory illnesses. The proposed study will be conducted at the Fima Lifshitz Metabolic Research Center, Department of Pediatrics, Universidade Federal Da Bahia, Salvador-Bahia, Brazil over a period of 18 months. This is a double-blind placebo-controlled trial involving the use of 2 types of micronutrient sprinkles in a group of 120 children who attend a day care center in Salvador, Bahia. They will be randomized into 2 groups of 60 children each. The intervention group will receive sprinkles containing zinc while the control group will receive micronutrient sprinkles without zinc. The primary outcome variables of interest are zinc status, stool zinc losses and diarrhea duration. Both groups of infants will be monitored at monthly intervals for an initial duration of 180 days for zinc status, diarrhea episodes, respiratory illness and growth. This study will allow for the establishment of a cohort of children who will be monitored in a micronutrient supplementation trial using sprinkles.

DETAILED DESCRIPTION:
The proposed study will be conducted at the Fima Lifshitz Metabolic Research Center, Department of Pediatrics, Universidade Federal Da Bahia, Salvador-Bahia, Brazil over a period of 18 months. This is a double-blind placebo-controlled trial involving the use of 2 types of micronutrient sprinkles in a group of 120 children who attend a day care center in Salvador, Bahia. They will be randomized into 2 groups of 60 children each. The intervention group will receive sprinkles containing zinc while the control group will receive micronutrient sprinkles without zinc. The primary outcome variables of interest are zinc status, stool zinc losses and diarrhea duration. Both groups of infants will be monitored at monthly intervals for an initial duration of 180 days for zinc status, diarrhea episodes, respiratory illness and growth. This study will allow for the establishment of a cohort of children who will be monitored in a micronutrient supplementation trial using sprinkles.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children attending day care

Exclusion Criteria:

* Chronic medical problems including sickle cell disease, congenital heart disease

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 143 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Conrad R Cole, MD, MPH, MSc, Principal Investigator — Emory University; Hugo Ribeiro Da Costa, MD, PhD, Principal Investigator — Universidade Federal da Bahia, Complexo Hospitalar Universitário Professor Edgar Santos, Centro de Pesquisa Fima Lifshitz, Salvador, Bahia, Brazil
Locations (1):
- Universidade Federal da Bahia, Complexo Hospitalar Universitário Professor Edgar Santos, Centro de Pesquisa Fima Lifshitz, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Derived] Imdad A, Rogner J, Sherwani RN, Sidhu J, Regan A, Haykal MR, Tsistinas O, Smith A, Chan XHS, Mayo-Wilson E, Bhutta ZA. Zinc supplementation for preventing mortality, morbidity, and growth failure in children aged 6 months to 12 years. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD009384. doi: 10.1002/14651858.CD009384.pub3. PMID 36994923

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy, 06 to 48 months old children attending a day care. They were randomized into two groups and received daily zinc micronutrient + - test group (sprinkles) or without zinc micronutrient only - control. Children were supplemented for 90 days
Groups:
- Micronutrient Sprinkles Without Zinc: Micronutrient sprinkles without zinc
  Micronutrient sprinkles without zinc : I packet of micronutrient sprinkles without zinc
- Micronutrient Sprinkles With Zinc: Micronutrient sprinkles with zinc gluconate
  Micronutrient Sprinkles with zinc : Daily dose of 1 packet of sprinkles
Period: Overall Study
Arm/Group | Micronutrient Sprinkles Without Zinc | Micronutrient Sprinkles With Zinc
Started | 68 | 75
Completed | 68 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Micronutrient Sprinkles Without Zinc | Micronutrient Sprinkles With Zinc | Total
Number analyzed (Participants) | 68 | 75 | 143
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 68 | 75 | 143
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 2.1 (2) | 2.2 (2) | 2.1 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 27 | 60
  Male | 35 | 48 | 83
Region of Enrollment [Number; unit: participants]
  Brazil | 68 | 75 | 143

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Children of Diarrhea Episodes
Description: Number of children with diarrhea divided by the number of children in the group
Time Frame: 6 months
Population: All children enrolled
Measure: Number; unit: percentage of participants
Arm/Group | Micronutrient Sprinkles Without Zinc | Micronutrient Sprinkles With Zinc
Number analyzed (Participants) | 68 | 75
percentage of participants | 19.1 | 14.7

2. Secondary Outcome: Proportion of Children With Respiratory Infections
Description: Number of children with respiratory infections divided by the total number of children in the group
Time Frame: 6 months
Population: All children enrolled
Measure: Number; unit: percentage of participants
Arm/Group | Micronutrient Sprinkles Without Zinc | Micronutrient Sprinkles With Zinc
Number analyzed (Participants) | 68 | 75
percentage of participants | 48.5 | 60

ADVERSE EVENTS:
Arm/Group | Micronutrient Sprinkles Without Zinc | Micronutrient Sprinkles With Zinc
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/75
Other Adverse Events (participants affected / at risk) | 0/68 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No